CLINICAL TRIAL: NCT00802724
Title: Classification-Directed Treatment of Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Linda Van Dillen, Associate Professor, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD047709-04; HD047709-04
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Low Back Pain
Keywords: low back pain; classification; spine
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Classification-directed treatment (Experimental): People in the Classification-directed treatment will be treated based on their direction-specific LBP classification. Treatment will consist of 3 primary components. The first component of treatment will be analysis and instruction in modification of the person's direction-specific alignment and movement strategies during symptomatic functional activities and activities in which the person uses similar strategies to those displayed with symptomatic functional activities. The second component is education about the principles of tissue injury and healing and the need to keep active. The third component is exercise prescription that consists of practice in performance of modified versions of the direction-specific impairment tests from the exam, with an emphasis on impairments that can be modified to eliminate symptoms.
  Interventions: Behavioral: Classification-directed treatment
- 2 Non-specific treatment (Active Comparator): People in the Non-specific treatment will be provided treatment that incorporates treatment commonly cited in the literature for people with chronic LBP. The first component of treatment will consist of training in functional activities based on biomechanical principles. The second component will include general education about low back pain. The third component is exercise prescription that is directed at improving the strength and flexibility of the trunk and limbs.
  Interventions: Behavioral: Non-specific treatment

INTERVENTIONS:
Behavioral: Classification-directed treatment — People in the Classification-directed treatment will be treated based on their direction-specific LBP classification. Treatment will consist of 3 primary components. The first component of treatment will be analysis and instruction in modification of the person's direction-specific alignment and movement strategies during symptomatic functional activities and activities in which the person uses similar strategies to those displayed with symptomatic functional activities. The second component is education about the principles of tissue injury and healing and the need to keep active. The third component is exercise prescription that consists of practice in performance of modified versions of the direction-specific impairment tests from the exam, with an emphasis on impairments that can be modified to eliminate symptoms.
  Arms: 1 Classification-directed treatment
Behavioral: Non-specific treatment — People in the Non-specific treatment will be provided treatment that incorporates treatment commonly cited in the literature for people with chronic LBP. The first component of treatment will consist of training in functional activities based on biomechanical principles. The second component will include general education about low back pain. The third component is exercise prescription that is directed at improving the strength and flexibility of the trunk and limbs.
  Arms: 2 Non-specific treatment

SUMMARY:
The primary purpose of this proposal is to conduct a prospective, randomized, controlled clinical trial to examine whether or not treatment based on a person's direction-specific, impairment-based LBP classification is more effective than Non-specific treatment in improving short- (6 weeks) and long-term (6 and 12 months) outcomes in people with chronic LBP. We hypothesize that treatment based on a person's direction-specific, impairment-based LBP classification (Classification-specific) will result in better outcomes than Non-specific treatment. Our approach to classification-directed treatment is based on the proposal that a person's LBP is the result of adopting direction-specific strategies of movement and alignment of the spine which then are used repeatedly during the person's everyday activities. The exposure of spine tissue to repeated loading in the same direction across a day is proposed to accelerate the accumulation of stress, microtrauma, and eventually LBP. We also hypothesize that until the factors contributing to the use of the direction-specific strategies of the spine are modified, the LBP problem will persist or recur. Identification of homogeneous subgroups of people with LBP will enhance 1) the power of clinical trials, 2) prognosis, and 3) the ability to identify mechanisms contributing to different LBP problems.

ELIGIBILITY:
Inclusion Criteria:

* People who report a history of chronic LBP for a minimum of 12 months,currently are experiencing LBP symptoms but not in an acute recurrence,
* Between 18 and 60 years of age,
* Able to stand and walk without assistance,
* Able to understand and read English,
* Able to understand and sign a consent form

Exclusion Criteria:

* Any structural spinal deformity including scoliosis, kyphosis, or stenosis,
* A spinal fracture or dislocation,
* Osteoporosis,
* Ankylosing spondylitis,
* Rheumatoid arthritis,
* Disc herniation,
* Serious spinal complications such as tumor or infection,
* Previous spinal surgery,
* Frank neurological loss, i.e., weakness and sensory loss,
* Pain or paresthesia below the knee,
* Etiology of LBP other than the lumbar spine, e.g., hip joint,
* History of neurologic disease which required hospitalization,
* Active treatment for cancer,
* History of unresolved cancer,
* Pregnancy,
* Magnified symptom behavior,
* Worker's compensation or disability case,
* In litigation for the LBP problem,
* Referral from a specialized pain clinic source,
* Spondylolisthesis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Modified Oswestry Disability Index for Low Back Pain (0-100%) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Functional limitation measure

SECONDARY OUTCOMES:
Kinematic measures of select movements and postures | Baseline, completion of treatment phase
  Impairment level measure
Numeric pain rating scale (0-10 points) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Impairment level measure
Medication use (yes, no) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Impairment level measure
Days of low back pain-related time off (number) | Baseline, 6 months after treatment phase, 12 months after treatment phase
  Impairment level measure; Question #5 from the Graded Chronic Pain Scale (Von Korff et al., Pain, 1990)
Baecke Habitual Activity Measure (3-15 points) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Impairment level measure
Fear Avoidance Beliefs Questionnaire Work subscale (0-42 points) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Impairment level measure
SF-36 Physical Functioning subscale (0-100%) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Disability level measure
SF-36 Role Functioning-Physical subscale (0-100%) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Disability level measure
SF-36 Bodily Pain subscale (0-100%) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Disability level measure
SF-36 General Health subscale (0-100%) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Disability level measure
SF-36 Vitality subscale (0-100%) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Disability level measure
SF-36 Social Functioning Subscale (0-100%) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Disability level measure
SF-36 Role Functioning subscale (0-100%) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Disability level measure
Fear Avoidance Beliefs Activity subscale (0-24 points) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Impairment level measure
SF-36 Role Functioning-Emotional subscale (0-100%) | Baseline, completion of treatment phase, 6 months, 12 months
  Disability level measure
SF-36 Mental Health subscale (0-100%) | Baseline, completion of treatment phase, 6 months after treatment phase,12 months after treatment phase
  Disability level measure
Adherence to exercise (0-100%) | Second treatment visit, completion of treatment phase, 6 months after treatment phase, 12 months after treatment phase
  Measure of the percentage of times the person reports adhering to performing the exercise as prescribed
Adherence to training in performance of functional activities (0-100%) | Second treatment visit, completion of treatment phase, 6 months post-treatment phase, 12 months post-treatment phase
  Measure of the percentage of times the person adhered to performing his/her functional activities as prescribed

OTHER OUTCOMES:
Satisfaction with care (15-75 points) | Completion of treatment phase
  Satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Van Dillen, P.T., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Holtzman G, Harris-Hayes M, Hoffman SL, Zou D, Edgeworth RA, Van Dillen LR. Clinical examination procedures to determine the effect of axial decompression on low back pain symptoms in people with chronic low back pain. J Orthop Sports Phys Ther. 2012 Feb;42(2):105-13. doi: 10.2519/jospt.2012.3724. Epub 2011 Oct 25. PMID 22027267
- [Background] Hoffman SL, Harris-Hayes M, Van Dillen LR. Differences in activity limitation between 2 low back pain subgroups based on the movement system impairment model. PM R. 2010 Dec;2(12):1113-8. doi: 10.1016/j.pmrj.2010.09.003. PMID 21145523
- [Background] Harris-Hayes M, Holtzman GW, Earley JA, Van Dillen LR. Development and preliminary reliability testing of an assessment of patient independence in performing a treatment program: standardized scenarios. J Rehabil Med. 2010 Mar;42(3):221-7. doi: 10.2340/16501977-0505. PMID 20411216
- [Background] Hoffman SL, Johnson MB, Zou D, Van Dillen LR. Differences in end-range lumbar flexion during slumped sitting and forward bending between low back pain subgroups and genders. Man Ther. 2012 Apr;17(2):157-63. doi: 10.1016/j.math.2011.12.007. Epub 2012 Jan 17. PMID 22261650
- [Background] Ravenna MM, Hoffman SL, Van Dillen LR. Low interrater reliability of examiners performing the prone instability test: a clinical test for lumbar shear instability. Arch Phys Med Rehabil. 2011 Jun;92(6):913-9. doi: 10.1016/j.apmr.2010.12.042. PMID 21621668
- [Background] Scholtes SA, Norton BJ, Lang CE, Van Dillen LR. The effect of within-session instruction on lumbopelvic motion during a lower limb movement in people with and people without low back pain. Man Ther. 2010 Oct;15(5):496-501. doi: 10.1016/j.math.2010.05.003. Epub 2010 Jun 2. PMID 20627798
- [Background] Harris-Hayes M, Van Dillen LR. The inter-tester reliability of physical therapists classifying low back pain problems based on the movement system impairment classification system. PM R. 2009 Feb;1(2):117-26. doi: 10.1016/j.pmrj.2008.08.001. Epub 2008 Dec 27. PMID 19627885
- [Background] Scholtes SA, Gombatto SP, Van Dillen LR. Differences in lumbopelvic motion between people with and people without low back pain during two lower limb movement tests. Clin Biomech (Bristol). 2009 Jan;24(1):7-12. doi: 10.1016/j.clinbiomech.2008.09.008. Epub 2008 Nov 5. PMID 18990474
- [Background] Henry SM, Van Dillen LR, Trombley AR, Dee JM, Bunn JY. Reliability of novice raters in using the movement system impairment approach to classify people with low back pain. Man Ther. 2013 Feb;18(1):35-40. doi: 10.1016/j.math.2012.06.008. Epub 2012 Jul 15. PMID 22796388
- [Result] Hoffman SL, Johnson MB, Zou D, Harris-Hayes M, Van Dillen LR. Effect of classification-specific treatment on lumbopelvic motion during hip rotation in people with low back pain. Man Ther. 2011 Aug;16(4):344-50. doi: 10.1016/j.math.2010.12.007. Epub 2011 Jan 20. PMID 21256073
- [Derived] Hoffman SL, Johnson MB, Zou D, Van Dillen LR. Sex differences in lumbopelvic movement patterns during hip medial rotation in people with chronic low back pain. Arch Phys Med Rehabil. 2011 Jul;92(7):1053-9. doi: 10.1016/j.apmr.2011.02.015. PMID 21704784